CLINICAL TRIAL: NCT03246100
Title: Centralized IIS-based Reminder/Recall to Increase Childhood Influenza Vaccination Rates, 2nd Trial in Colorado
Brief Title: Centralized IIS-based Reminder/Recall to Increase Childhood Influenza Vaccination Rates_2nd Trial in Colorado
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 15-0570_2
Record Dates: First submitted 2017-08-07; First posted 2017-08-11 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Reminder Systems; Influenza Vaccines
Keywords: centralized reminder/recall; influenza vaccine reminders; childhood influenza vaccines
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Patients will be randomized within practices to one of 3 arms:
  1. Standard of care control
  2. Autodialer (3 reminders)- with brief education message + practice name + practice phone # (see autodialer scripts)
  3. Mailed reminder (3 reminders)-- with brief education message + practice name + practice phone # (see postcards)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): These patients will receive no reminders from the health department and will receive usual care.
- Autodialer R/R (Experimental): Autodialer calls (up to 3 reminders)- with brief education message + practice name + practice phone #
  Interventions: Behavioral: Reminders
- Mail R/R (Experimental): Mailed reminder (up to 3 reminders)-- with brief education message + practice name + practice phone #
  Interventions: Behavioral: Reminders

INTERVENTIONS:
Behavioral: Reminders — Reminders are sent either through autodial or postcards reminding patients to get flu vaccine.
  Arms: Autodialer R/R; Mail R/R

SUMMARY:
This study is the second trial related to ClinicalTrials.gov ID: NCT02761551. There are slight changes to methods and a different cohort will be used, thus justifying a 2nd ClinicalTrials.gov submission. This trial is taking place in New York State (not NYC) and in Colorado. Each state has it's own ClinicalTrials.gov submission.

Despite U.S. guidelines for influenza vaccination of all children starting at age 6 months, only about half of children are vaccinated annually leading to substantial influenza disease in children and spread of disease to adults. A major barrier is that families are not reminded about the need for their children to receive influenza vaccination. The investigators will evaluate the impact of patient reminder/recall (R/R) performed by state immunization information systems to improve influenza vaccination rates by using three clinical trials in two states. The investigators will assess effectiveness and cost-effectiveness of: 1) autodialer reminder/recall versus 2) postcard reminder/recall versus 3) usual care (no R/R) on improving influenza vaccination rates.

The investigators will disseminate the state immunization information system based reminder/recall system to all states for use for both seasonal and pandemic influenza vaccinations with the goal of lowering influenza morbidity.

DETAILED DESCRIPTION:
Annual epidemics of seasonal influenza cause substantial morbidity and mortality in the U.S. with high rates of hospitalizations, emergency department and outpatient visits, and medical costs. Children experience significant morbidity from influenza, and also play a critical role in spreading infection to adults. Since 2010, the Advisory Committee on Immunization Practices (ACIP) has recommended influenza vaccination for all children >6 months of age. However, vaccination rates remain very low-- only 56% of children 2-17 years are vaccinated. Low rates are a concern for both seasonal influenza and in preparation for pandemic influenza. One of the nationally recommended strategies for raising childhood influenza vaccination rates is to use parent reminder/recall (R/R) by phone or mail, which can raise rates by up to 20 percentage points. However, less than 16% of primary care practices use R/R despite many studies showing its effectiveness.

Statewide immunization information systems (IISs) now exist in all states to track childhood vaccinations, but they have not been used for R/R for influenza vaccine because of the lack of evidence for its effectiveness and lack of a template for IIS-based R/R. The investigators have united two leading immunization research groups (Denver, CO and Rochester, NY) to assess the impact of centralized IIS-based influenza vaccine R/R, and to evaluate the effect of two types of R/R (autodial v. mail R/R) over usual care. The investigators will also develop tools to aid other states in creating efficient IIS R/R systems for seasonal and possible pandemic influenza outbreaks.

In Colorado, evaluate the impact of (a) autodialer reminders and (b) mailed messages versus standard-of-care control on raising influenza vaccination rates among children 6m-17 years of age.

The investigators propose a 3-arm RCT study design with the following study arms:

1. Standard of care control
2. Autodialer (3 reminders)- with brief education message + practice name + practice phone #
3. Mailed reminder (3 reminders)-- with brief education message + practice name + practice phone #

ELIGIBILITY:
Inclusion Criteria:

* have record in Colorado Immunization Information System
* from 6 months through 17 years of age
* have not received an influenza vaccine by start of trial
* must be affiliated with one of our 42 randomly selected primary care practices in Colorado

Exclusion Criteria:

* those without a record
* received an influenza vaccine post 9/1/2017
* not affiliated with an eligible study

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25531 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Receipt of at least 1 influenza vaccine according to immunization records in the Immunization Information System (IIS) records in each state | 6 months
  Based on our prior studies, we currently plan to send up to 3 autodialer or postcards (based on randomization arm) reminders, spaced every 5 weeks, beginning in early October, and ending mid-December 2017. Outcomes are assessed at 6 months using IIS data.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kempe, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate results will be prepared for publications at the end of the trial.

REFERENCES:
- [Derived] Szilagyi PG, Albertin CS, Saville AW, Valderrama R, Breck A, Helmkamp L, Zhou X, Vangala S, Dickinson LM, Tseng CH, Campbell JD, Whittington MD, Roth H, Rand CM, Humiston SG, Hoefer D, Kempe A. Effect of State Immunization Information System Based Reminder/Recall for Influenza Vaccinations: A Randomized Trial of Autodialer, Text, and Mailed Messages. J Pediatr. 2020 Jun;221:123-131.e4. doi: 10.1016/j.jpeds.2020.02.020. PMID 32446470